CLINICAL TRIAL: NCT05981066
Title: An Open, Single-center, Multiple-dose, Dose-increasing and Dose-expanding Clinical Study to Observe and Evaluate the Safety, Tolerance, Immunokinetics and Preliminary Effectiveness of ABOR2014 Injection (IPM511) in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: A Clinical Study of mRNA Vaccine (ABOR2014/IPM511) in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J-23PJ957
Record Dates: First submitted 2023-07-05; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: mRNA vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPM511 monotherapy (Experimental): 3+3 dose excalation. Paticipants will receive two cycle (QWX4 per cycle) IPM511 injection，I.M injection
  Interventions: Drug: Neoantigen vaccine, I.M injection

INTERVENTIONS:
Drug: Neoantigen vaccine, I.M injection — Patients will receive a fixed applicable dose of ABOR2014(IPM511) administered.

SUMMARY:
This is an open label, single-site, investigator-initiated trial designed to evaluate the safety, tolerability and preliminary efficacy of ABOR2014(IPM511) injection in relapsed/ refactory HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand and voluntarily sign the informed consent form;
2. Male or female subjects ≥ 18 years old;
3. Patients with pathological or cytological evidence of locally advanced or hepatocellular carcinoma, who have failed or are intolerant of previous standard treatments;
4. At least one measurable lesion judged according to the RECIST version 1.1 standard.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 (inclusive);
6. Life expectancy ≥ 12 weeks;
7. HLA typing: A-02;
8. Laboratory tests at screening shall meet the following requirements:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
   * Platelet count (PLT) ≥ 90 × 10^9/L;
   * Hemoglobin (Hb) ≥ 90 g/L;
   * Total bilirubin (TBIL) ≤ 3 × ULN;
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × ULN;
   * Blood creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (calculated based on Cockcroft-Gault formula) ≥ 45 mL/min;
   * International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN;
   * QTc interval (calculated based on Fridericia's formula) ≤ 450 ms for males and ≤ 470 ms for females;
9. For subjects with hepatitis B-related primary hepatocellular carcinoma (HBV-HCC) or hepatitis C-related primary hepatocellular carcinoma (HCV-HCC), those who are with the following conditions are eligible to be enrolled:

   * HBV-HCC: resolved HBV infection with concomitant antiviral therapy;
   * HCV-HCC: resolved or active HCV infection , where concomitant antiviral therapy may be given for active HCV infection;

9. For patients of childbearing potential (male or female), effective contraceptive measures shall be taken during the study treatment and within 3 months after the last dose. For women of childbearing potential, a negative serum/urine HCG test result within 7 days prior to study enrollment shall be provided.

Exclusion Criteria:

1. Known allergy to any of the components of the investigational product;
2. History of topical treatment with mRNA products or treatment with mRNA vaccines;
3. Patients with a history of major operations within 4 weeks before the first dose, have a plan of major operations during the study (at the investigator's discretion);
4. History of anti-tumor therapies within 4 weeks before the first dose;
5. History of receiving immunosuppressive drugs within 4 weeks before the first dose, except for corticosteroid nasal sprays, inhalants, and systemic prednisone at a dose of ≤ 10 mg/day or similar drugs at equivalent doses;
6. History of organ transplant, bone marrow transplant, or hematopoietic stem cell transplant;
7. History of hemorrhagic diseases such as anaphylactoid purpura, Haemophilia and aplastic anemia;
8. History of live attenuated vaccines within 30 days before the first dose;
9. Central nervous system (CNS) metastases that are symptomatic, untreated, or require continuous treatment;
10. Toxicological events (except alopecia and pigmentation) have not recovered to baseline or NCI-CTCAE v5.0 grade 0-1 after prior anti-tumor therapies;
11. History of autoimmune disorders;
12. History of immediate hypersensitivity, eczema that cannot be controlled by topical corticosteroids, or asthma;
13. Uncontrollable concomitant diseases;
14. Active infections currently requiring systemic anti-infective therapy; active pulmonary tuberculosis;
15. Known history of human immunodeficiency virus (HIV) positive or treponema pallidum positive;
16. Patients with other conditions that are not suitable for participation in the study at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) | up to 12 months
  AE assessed according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Clinically significant abnormal changes in vital signs | up to 12 months
Clinically significant abnormal changes in laboratory tests | up to 12 months

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of IPM511 | up to 12 months
Time of Maximum Plasma Concentration [Tmax] of IPM511 | up to 12 months
Half-time of Plasma Concentration [T1/2] of IPM511 | up to 12 months
Antigen-specific T-cell responses in peripheral blood | up to 12 months
  Detected by Tetramer or TCRseq or Enzyme-linked Immunospot Assay(ELISPOT)
Change of Circulating tumor DNA (ctDNA) status (every 6 weeks) | up to 12 months
Objective Response Rate, ORR | up to 12 months
  ORR is Defined as the number of patients with a complete response (CR) or partial response(PR) .
Duration of Response, DoR | up to 12 months
  DoR is defined as time from first tumor response(partial or complete) until either radiogical disease progress, clinical/ symptomatic disease progression or death (whichever is sooner).
Progress Free Survival, PFS | up to 12 months
  PFS is defined as time between the date of first dose of IPM511 and the date either radiogical disease progress, clinical/ symptomatic disease progression or death (whichever is sooner).
Overall Survival, OS | up to 12 months
  OS is defined as time between the date of first dose of IPM511 and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No